CLINICAL TRIAL: NCT02259491
Title: Honey Dressings for Local Wound Care of Split Thickness Skin Graft and Free Tissue Transfer Donor Sites: A Prospective, Randomized, Controlled Trial.
Brief Title: Manuka Honey for Wound Care
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 13-1507
Record Dates: First submitted 2014-10-01; First posted 2014-10-08 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2018-02

CONDITIONS: Wound Healing
Keywords: Wound Healing; Honey; Skin Grafts; Free tissue transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manuka Honey Dressing (Experimental): Patient receive manuka honey dressings on skin graft and free flap donor sites
  Interventions: Other: Manuka Honey Dressing
- Tegaderm and xeroform gauze (No Intervention): Patient receive standard wound care on skin graft and free flap donor sites which includes a tegaderm over the STSG site and xeroform gauze covered with dry gauze, kerlex and a cast for the STSG recipient site

INTERVENTIONS:
Other: Manuka Honey Dressing — After surgical resection and reconstruction the skin graft donor site (thigh) and the free flap donor site will be dressed with Medihoney surgical dressings. More specifically, a dressing of appropriate size will be applied to the anterior thigh and covered with tegaderm. For the STSG recipient site a Medihoney dressing will cover the skin graft, followed by dry gauze, kerlex and a cast.
  Other Names: Medihoney; Calcium algninate dressings; Dermasciences
  Arms: Manuka Honey Dressing

SUMMARY:
Since antiquity, honey has been recognized for its healing properties. Literature about the use of medicinal honey for wound care dates back centuries with recent data suggesting its use in patients suffering from burns or pressure ulcers. Research has shown Manuka honey (Leptospermum scoparium) to have significant immune benefits and the ability to influence all phases of wound healing: inflammation, proliferation and remodeling. In addition, numerous clinical studies have identified positive benefits for wound healing. However, there is a lack of prospective, randomized controlled data on the use of honey as a medicinal agent in local wound care and scar healing.

In order to better understand Manuka Honey's ability to aid in healing, the investigators are conducting a randomized, controlled, single-blinded study of patients undergoing reconstructive surgery. This project uses split thickness skin graft and free tissue transfer donor sites as standard wound models to compare the effects of Manuka Honey versus standard wound care therapies. Through the use of standard wound model and objective measurement tools, the investigators hope to better elucidate any benefits of this novel wound care 'technology.'

DETAILED DESCRIPTION:
Free tissue transfer (FTT) and split-thickness skin grafting (STSG) are important aspects of head and neck reconstruction. The radial forearm skin flap and fibula osteocutaneous flap are commonly used in head and neck reconstruction. After harvest, closure of these donor sites often requires split thickness skin grafting. The grafting is usually done from the thigh. The grafted free flap donor site along with the STSG donor site is often the source of significant post-operative pain and complications including delayed wound healing, graft loss and infection. There is no consensus in the literature on the best care for these donor sites with surgeons employing a wide variety of surgical dressings for local wound care. There is literature dating back centuries on the use of medicinal honey for wound care, with recent data suggesting its use in patients suffering from burns or pressure ulcers. However, there is a lack of prospective, randomized controlled data on the use of honey as a medicinal agent in local wound care.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 undergoing reconstructive surgery with FTT and/or STSG

Exclusion Criteria:

* All patients under the age of 18
* Any patients with documented honey allergy
* Patients with documented collagen vascular diseases
* Patients with documented coagulopathy
* Patients with history of prior skin grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Scar Scale | up to 7 days
  Physician assessment of scar by Modified Vancouver Scar Scale

SECONDARY OUTCOMES:
Pain scores | up to 7 days
  Assessed by standardized and validated post-operative pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rosenberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States